CLINICAL TRIAL: NCT06868264
Title: Phase 3, Randomized, Controlled, Open-label Study to Compare the Efficacy and Safety of Bemnifosbuvir-Ruzasvir Fixed-dose Combination (BEM/RZR FDC) Versus Sofosbuvir-Velpatasvir Fixed-dose Combination (SOF/VEL FDC) in Subjects With Chronic Hepatitis C Virus (HCV) Infection
Brief Title: C-BEYOND: Efficacy and Safety of BEM/RZR vs. SOF/VEL in Subjects With Chronic HCV
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT-01B-007
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: HEPATITIS C VIRUS CHRONIC INFECTION
MeSH Terms: interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bemnifosbuvir-Ruzasvir (BEM/RZR) (Experimental)
  Interventions: Drug: Bemnifosbuvir-Ruzasvir (BEM/RZR)
- Sofosbuvir-Velpatasvir (SOF/VEL) (Active Comparator)
  Interventions: Drug: Sofosbuvir-Velpatasvir (SOF/VEL)

INTERVENTIONS:
Drug: Bemnifosbuvir-Ruzasvir (BEM/RZR) — BEM/RZR Fixed-dose Combination (FDC) tablets administered orally once daily for a total of 8 weeks (in those without cirrhosis) or 12 weeks (in those with compensated cirrhosis)
  Arms: Bemnifosbuvir-Ruzasvir (BEM/RZR)
Drug: Sofosbuvir-Velpatasvir (SOF/VEL) — SOF/VEL Fixed-dose Combination (FDC) tablets administered orally once daily for a total of 12 weeks
  Arms: Sofosbuvir-Velpatasvir (SOF/VEL)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of BEM/RZR to SOF/VEL in adults with chronic HCV.

ELIGIBILITY:
Key Inclusion Criteria:

* Use of adequate contraception for females of childbearing potential
* Must be direct-acting antiviral (DAA)-treatment-naïve (never exposed to an approved or experimental DAA for HCV)
* Documented medical history compatible with chronic HCV
* Either no liver cirrhosis or with compensated liver cirrhosis
* If HIV-1-positive, must meet the following 2 criteria:

  1. Antiretroviral (ARV) regimen for >8 weeks prior to screening visit, with CD4 T-cell count >200 cells/mm3 and plasma HIV-1 RNA <LLOQ
  2. Suitable ARV treatment and not taking any contraindicated medications

Key Exclusion Criteria:

* Pregnant or breastfeeding
* Co-infected with hepatitis B virus
* Abuse of alcohol and/or illicit drug use that could interfere with adherence to study requirements as judged by the investigator
* Requirement of any prohibited medications
* Use of other investigational drugs within 30 days of dosing
* History or signs of decompensated liver disease (decompensated cirrhosis)
* History of hepatocellular carcinoma (HCC)
* Any other clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving HCV RNA less than the lower limit of quantitation (LLOQ) at study week 24. | Day 1 through Week 24

SECONDARY OUTCOMES:
Proportion of subjects achieving HCV RNA < LLOQ 12 weeks after the last dose of study drugs. | Day 1 through 12 weeks after the end of treatment
Proportion of subjects experiencing virologic failure. | Day 1 through Week 24

CONTACTS AND LOCATIONS:
Locations (95):
- United States (87):
  - Atea Study Site, Birmingham, Alabama
  - Atea Study Site, Dothan, Alabama
  - Atea Study Site, Chandler, Arizona
  - Atea Study Site, Flagstaff, Arizona
  - Atea Study Site, Mesa, Arizona
  - Atea Study Site, Phoenix, Arizona
  - Atea Study Site, Tucson, Arizona
  - Atea Study Site, Little Rock, Arkansas
  - Atea Study Site, Bakersfield, California
  - Atea Study Site, Coronado, California
  - Atea Study Site, Escondido, California
  - Atea Study Site, Fresno, California
  - Atea Study Site, Long Beach, California
  - Atea Study Site, Los Angeles, California
  - Atea Study Site, Orange, California
  - Atea Study Site, Pasadena, California
  - Atea Study Site, Sacramento, California
  - Atea Study Site, Torrance, California
  - Atea Study Site, Valencia, California
  - Atea Study Site, Colorado Springs, Colorado
  - Atea Study Site, Washington D.C., District of Columbia
  - Atea Study Site, Coral Gables, Florida
  - Atea Study Site, DeLand, Florida
  - Atea Study Site, Fort Lauderdale, Florida
  - Atea Study Site, Ft. Pierce, Florida
  - Atea Study Site, Gainesville, Florida
  - Atea Study Site, Inverness, Florida
  - Atea Study Site, Jupiter, Florida
  - Atea Study Site, Lauderdale Lakes, Florida
  - Atea Study Site, Maitland, Florida
  - Atea Study Site, Miami, Florida
  - Atea Study Site, Miami Lakes, Florida
  - Atea Study Site, Orlando, Florida
  - Atea Study Site, Pembroke Pines, Florida
  - Atea Study Site, Sarasota, Florida
  - Atea Study Site, West Palm Beach, Florida
  - Atea Study Site, Macon, Georgia
  - Atea Study Site, Marietta, Georgia
  - Atea Study Site, Chicago, Illinois
  - Atea Study Site, New Albany, Indiana
  - Atea Study Site, Fairway, Kansas
  - Atea Study Site, Topeka, Kansas
  - Atea Study Site, Louisville, Kentucky
  - Atea Study Site, New Iberia, Louisiana
  - Atea Study Site, New Orleans, Louisiana
  - Atea Study Site, Baltimore, Maryland
  - Atea Study Site, Boston, Massachusetts
  - Atea Study Site, Springfield, Massachusetts
  - Atea Study Site, Worcester, Massachusetts
  - Atea Study Site, Detroit, Michigan
  - Atea Study Site, Grosse Pointe Woods, Michigan
  - Atea Study Site, Novi, Michigan
  - Atea Study Site, Wyoming, Michigan
  - Atea Study Site, Tupelo, Mississippi
  - Atea Study Site, Camden, New Jersey
  - Atea Study Site, Hackensack, New Jersey
  - Atea Study Site, Hillsborough, New Jersey
  - Atea Study Site, Newark, New Jersey
  - Atea Study Site, Brooklyn, New York
  - Atea Study Site, New York, New York
  - Atea Study Site, Yonkers, New York
  - Atea Study Site, Asheville, North Carolina
  - Atea Study Site, Charlotte, North Carolina
  - Atea Study Site, Fayetteville, North Carolina
  - Atea Study Site, Beavercreek, Ohio
  - Atea Study Site, Cincinnati, Ohio
  - Atea Study Site, Tulsa, Oklahoma
  - Atea Study Site, Allentown, Pennsylvania
  - Atea Study Site, DuBois, Pennsylvania
  - Atea Study Site, Philadelphia, Pennsylvania
  - Atea Study Site, Charleston, South Carolina
  - Atea Study Site, Chattanooga, Tennessee
  - Atea Study Site, Cordova, Tennessee
  - Atea Study Site, Jackson, Tennessee
  - Atea Study Site, Arlington, Texas
  - Atea Study Site, Dallas, Texas
  - Atea Study Site, Denison, Texas
  - Atea Study Site, Houston, Texas
  - Atea Study Site, Plano, Texas
  - Atea Study Site, San Antonio, Texas
  - Atea Study Site, Temple, Texas
  - Atea Study Site, Waco, Texas
  - Atea Study Site, Ogden, Utah
  - Atea Study Site, Chesapeake, Virginia
  - Atea Study Site, Norfolk, Virginia
  - Atea Study Site, Richmond, Virginia
  - Atea Study Site, Seattle, Washington
- Canada (8):
  - Atea Study Site, Vancouver, British Columbia
  - Atea Study Site, Moncton, New Brunswick
  - Atea Study Site, St. John's, Newfoundland and Labrador
  - Atea Study Site, Brampton, Ontario
  - Atea Study Site, Ottawa, Ontario
  - Atea Study Site, Toronto, Ontario
  - Atea Study Site, Montreal, Quebec
  - Atea Study Site, Québec, Quebec